CLINICAL TRIAL: NCT05340036
Title: Skeletal Stability of Le Fort I Osteotomy Using Patient-specific Osteosynthesis Compared to Mini-plate Fixation for Patients With Dentofacial Disharmony. A Randomized Controlled Clinical Trial
Brief Title: Skeletal Stability of Le Fort I Osteotomy Using Patient-specific Osteosynthesis Compared to Mini-plate Fixation for Patients With Dentofacial Disharmony
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hassan Fahmy Hassan Alnimr (Other)
Responsible Party: Sponsor-Investigator, Hassan Fahmy Hassan Alnimr, Principal Investigator, Cairo University
Organization: Cairo University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: OMFS 3 3 7
Record Dates: First submitted 2022-04-04; First posted 2022-04-21 (Actual); Last update posted 2022-06-01 (Actual); Status verified 2022-05

CONDITIONS: Dentofacial Deformities
Keywords: orthognathic surgery; virtual planning; customized titanium plates; cutting guides; CAD/CAM
MeSH Terms: conditions — Dentofacial Deformities

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: Due to the nature of the intervention, therapists cannot be blinded to allocation, but are strongly instructed not to disclose the allocation status to the participant at the follow up assessments. Mrs. Esraa will feed data into the computer in separate datasheets so that the assessors can analyze data without having access to information about the allocation and the procedure.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group I (Conventional plates) (Active Comparator): Digital intermediate and final interocclusal wafer splints will be designed to guide the maxilla and mandible in the desired position using CAD software (3-matic 11.0; Materialise NV, Leuven, Belgium).
  The designed splints will be then exported in stereolithography (STL) file format to the additive CAM machine (FORMIGA P 110 printer; EOS e-manufacturing solutions, Munich, Germany) and manufactured in white polyamide (PA2200; EOS e-manufacturing solutions, Munich, Germany) using fused deposition modelling (FDM) technology.The splints will be cold sterilized by overnight immersion in 2% glutaraldehyde.
  2.0 conventional mini plates will be used for fixation of maxilla and mandible in the new position.
  Interventions: Procedure: Bimaxillary orthognathic surgery using conventional plates
- Group II (Patient specific plates) (Experimental): The cutting guides will be designed on the maxilla and mandible to orient the osteotomy and mark reference holes to be used later for the repositioning/ fixation plate, using CAD software.
  The designed guide will be then exported in stereolithography (STL) file format to the additive CAM machine and manufactured in white polyamide using fused deposition modelling (FDM) technology. No finishing or polishing was done in order to maintain accuracy. The guides will be cold sterilized by overnight immersion in 2% glutaraldehyde.
  The patient-specific osteosynthesis plates will be designed to fix the maxilla and mandible in the desired position making use of the previously established reference holes. The designed plates will be exported in STL file format to be manufactured in grade 5 titanium alloy utilizing selective laser sintering (SLS) technology on an additive CAM machine.
  Interventions: Procedure: Bimaxillary orthognathic surgery using patient specific plates

INTERVENTIONS:
Procedure: Bimaxillary orthognathic surgery using conventional plates — le fort I osteotomy will carried out in the classic way guided by the classic landmarks (maxillary roots apices) as described by Wassmund.
  Complete separation of the maxillary segment using chisels and mallets in regular fashion.
  Reposition maxilla using the interocclusal wafer while mandible is gently positioned to centric relation position.
  Mandible is maintained in place until fixation of the maxilla with plates and screws takes place.
  Complete separation of the mandibular segment using chisels and mallets in regular fashion.
  Repositioning of mandible using the final interocclusal wafer while condylar segment is gently positioned to centric relation position.
  Fixation of mandibular segments with plates and/or screws in regular fashion.
  Incision was closed with 4-0 resorbable sutures in a continuous running fashion.
  Arms: Group I (Conventional plates)
Procedure: Bimaxillary orthognathic surgery using patient specific plates — The cutting guide of the maxilla will be placed onto the exposed bony surface and manipulated to the best fit.
  Then, the guide will be fixed using four 2.0-mm screws to avoid any mobilization during drilling of the reference holes. Sixteen reference holes will be established using the cutting guide; eight on each side.
  Then, a reciprocating saw will be used to perform the planned Le Fort I osteotomy. After adequate maxillary mobilization and removal of bony interferences, the maxilla will be repositioned using the patient-specific osteosynthesis material guided by the previously established reference holes and fixed using 2.0-mm screws.
  Then, the mandibular cutting guide will be fixed in the same manner and bilateral sagittal split osteotomy will be carried out.
  After adequate mobilization, the mandible will be repositioned by the patient-specific osteosynthesis material using the reference holes made by cutting guide and fixed using 2.0-mm screws.
  Arms: Group II (Patient specific plates)

SUMMARY:
The aim of the study is to evaluate the Skeletal stability of Le Fort I osteotomy using patient-specific osteosynthesis compared to Mini-plate fixation for patients with skeletal class III malocclusion.

DETAILED DESCRIPTION:
postsurgical relapse is one of the most common observations that have been reported after fixation of Le Fort I osteotomy cases.

Fixation systems with plates and screws are used in oral maxillofacial surgery for the treatment of facial fractures and orthognathic surgery cases. Although they have been used for decades and have become the standard treatment, the materials used in these systems may fail due to excess loading and other causal factors during the surgical procedure, including failure in plate adaptation and fixation to bone, material design, fabrication, and degree of purity of the plate material.

In the fixation system, non-customized plates of standard size are used, and are bent to adapt them to the distances required for planning orthognathic surgeries. Therefore, mandatory use of larger plates than those programmed for use in surgeries is required so that they can be bent to enable insertion. Moreover, there are variations in the number of screws required to retain the plates to enable better fixation. The folds of non-customized plates generate stresses that are minimized when using customized plates, because these plates are fabricated individually, with predetermined sizes for each patient.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with skeletal class III malocclusion planned for traditional Orthognathic Approach and requiring bimaxillary orthognathic surgeries in which there will be Le Fort I osteotomy with maxillary advancement ranging from 2mm to 5 mm in addition to mandibular setback.
2. Patients with no signs or symptoms of active TMDs.
3. Highly motivated patients.

Exclusion Criteria:

1. Patients who refused to be included in the research.
2. Patients with systemic diseases that may hinder the normal healing process or render the patient not fitting for general anaesthesia.
3. Patients with intra-bony lesions or infections that may retard the osteotomy healing.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2022-05-26 (Actual); Primary Completion 2023-11 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Skeletal relapse of Le Fort I osteotomy | Linear deviations between immediate postoperative and 12 months postoperative position
  Skeletal relapse will be assessed through measuring Linear deviations (DT) between the immediate postoperative (T1) and the 12 months postoperative position (T2) in Mimics 19.0 software using hard tissue reference points (A point, Anterior nasal spine, posterior nasal spine, Incisive foramen, Right side Greater palatine foramen, Left side Greater palatine foramen) in relation to three reference planes (Frankfort horizontal plane (FHP), coronal plane, and mid-facial plane (MFP)). Measurements from the reference points to the FHP indicated vertical deviation, to the coronal plane indicated anteroposterior deviation, and to the MFP indicated mediolateral deviation. measurements will be in millimeters.

CONTACTS AND LOCATIONS:
Overall Officials: Hassan Alnimr, Principal Investigator — Cairo University
Locations (1):
- Faculty of Dentistry, Cairo University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be available to other researchers.

REFERENCES:
- [Background] Ohba S, Nakao N, Nakatani Y, Yoshimura H, Minamizato T, Kawasaki T, Yoshida N, Sano K, Asahina I. Effects of Vertical Movement of the Anterior Nasal Spine on the Maxillary Stability After LeFort I Osteotomy for Pitch Correction. J Craniofac Surg. 2015 Sep;26(6):e481-5. doi: 10.1097/SCS.0000000000001968. PMID 26267571
- [Background] Lee CC, Xhori O, Tannyhill RJ, Kaban LB, Peacock ZS. Variables associated with stability after Le Fort I osteotomy for skeletal class III malocclusion. Int J Oral Maxillofac Surg. 2021 Sep;50(9):1203-1209. doi: 10.1016/j.ijom.2021.02.004. Epub 2021 Feb 28. PMID 33658151
- [Background] Wangsrimongkol B, Flores RL, Staffenberg DA, Rodriguez ED, Shetye PR. Skeletal and Dental Correction and Stability Following LeFort I Advancement in Patients With Cleft Lip and Palate With Mild, Moderate, and Severe Maxillary Hypoplasia. Cleft Palate Craniofac J. 2022 Jan;59(1):98-109. doi: 10.1177/1055665621996108. Epub 2021 Mar 15. PMID 33722088
- [Background] Ramos VF, Pinto LAPF, Basting RT. Force and deformation stresses in customized and non-customized plates during simulation of advancement genioplasty. J Craniomaxillofac Surg. 2017 Nov;45(11):1820-1827. doi: 10.1016/j.jcms.2017.08.021. Epub 2017 Aug 31. PMID 28935483
- [Background] Stokbro K, Borg SW, Andersen MO, Thygesen T. Patient-specific 3D printed plates improve stability of Le Fort 1 osteotomies in vitro. J Craniomaxillofac Surg. 2019 Mar;47(3):394-399. doi: 10.1016/j.jcms.2018.12.015. Epub 2019 Jan 3. PMID 30661925
- [Background] Kotaniemi KVM, Heliovaara A, Kotaniemi M, Stoor P, Leikola J, Palotie T, Suojanen J. Comparison of postoperative skeletal stability of maxillary segments after Le Fort I osteotomy, using patient-specific implant versus mini-plate fixation. J Craniomaxillofac Surg. 2019 Jul;47(7):1020-1030. doi: 10.1016/j.jcms.2019.04.003. Epub 2019 Apr 27. PMID 31085061
- [Background] Buijs GJ, van Bakelen NB, Jansma J, de Visscher JG, Hoppenreijs TJ, Bergsma JE, Stegenga B, Bos RR. A randomized clinical trial of biodegradable and titanium fixation systems in maxillofacial surgery. J Dent Res. 2012 Mar;91(3):299-304. doi: 10.1177/0022034511434353. Epub 2012 Jan 23. PMID 22269272
- [Background] Larsen AJ, Van Sickels JE, Thrash WJ. Postsurgical maxillary movement: a comparison study of bone plate and screw versus wire osseous fixation. Am J Orthod Dentofacial Orthop. 1989 Apr;95(4):334-43. doi: 10.1016/0889-5406(89)90167-4. PMID 2705414
- [Background] Park JH, Kim M, Kim SY, Jung HD, Jung YS. Three-dimensional analysis of maxillary stability after Le Fort I osteotomy using hydroxyapatite/poly-L-lactide plate. J Craniomaxillofac Surg. 2016 Apr;44(4):421-6. doi: 10.1016/j.jcms.2016.01.011. Epub 2016 Jan 19. PMID 26880012
- [Background] Hanafy M, Akoush Y, Abou-ElFetouh A, Mounir RM. Precision of orthognathic digital plan transfer using patient-specific cutting guides and osteosynthesis versus mixed analogue-digitally planned surgery: a randomized controlled clinical trial. Int J Oral Maxillofac Surg. 2020 Jan;49(1):62-68. doi: 10.1016/j.ijom.2019.06.023. Epub 2019 Jun 29. PMID 31262680
- [Background] Al-Delayme R, Al-Khen M, Hamdoon Z, Jerjes W. Skeletal and dental relapses after skeletal class III deformity correction surgery: single-jaw versus double-jaw procedures. Oral Surg Oral Med Oral Pathol Oral Radiol. 2013 Apr;115(4):466-72. doi: 10.1016/j.oooo.2012.08.443. Epub 2012 Nov 22. PMID 23177758
- [Background] Dupont WD, Plummer WD Jr. Power and sample size calculations. A review and computer program. Control Clin Trials. 1990 Apr;11(2):116-28. doi: 10.1016/0197-2456(90)90005-m. PMID 2161310
- [Background] Suojanen J, Leikola J, Stoor P. The use of patient-specific implants in orthognathic surgery: A series of 32 maxillary osteotomy patients. J Craniomaxillofac Surg. 2016 Dec;44(12):1913-1916. doi: 10.1016/j.jcms.2016.09.008. Epub 2016 Sep 23. PMID 27769722